CLINICAL TRIAL: NCT06154499
Title: Archive Prostate. Observational Study of Patients Who Underwent Radical Prostatectomy Surgery. Long-term Evaluation of the Course of Prostate Cancer Associated With Quality of Life, Post-surgery Treatments and Occurrence of Any Disease Recurrence
Brief Title: Archive Prostate. Observational Study of Patients Who Underwent Radical Prostatectomy Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Montorsi, Professor, IRCCS San Raffaele
Other Study IDs: 2004- Prostata
Record Dates: First submitted 2023-10-13; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred to the Urology Department who need to undergo radical prostatectomy surgery
  Interventions: Procedure: Radical prostatectomy

INTERVENTIONS:
Procedure: Radical prostatectomy — Radical Prostatectomy: surgery to remove the prostate gland and seminal vesicles (and sometimes nearby lymph nodes) after a prostate cancer diagnosis

SUMMARY:
This is a single-center, observational, prospective study on quality of life and disease status of patients who underwent radical prostatectomy. Data related to clinical conditions (oncological, psychological, sexual and quality of life) of these patients are collected in a database.

DETAILED DESCRIPTION:
A database was created with the intention of collecting data related to patients with diagnosis of prostate cancer who underwent radical prostatectomy.

Anamnesis, surgery, histological report and hospitalization data are collected for patients who underwent radical prostatectomy.

Each patient will be followed for 10 years from the date of radical prostatectomy surgery.

Each patient will receive a questionnaire before radical prostatectomy in order to evaluate the quality of life (urinary continence, erectile function and psycho-physical wellbeing). A follow up questionnaire will be collected after surgery in order to analyze the predictive factors of the disease, clinical progression and to obtain health benefits for the patients involved and for future patients with the same tipe of cancer, improving the scientific knowledge of the pathology and implementing new strategies for diagnosis and therapy and evaluating the epidemiologic changes of prostate cancer. Tha data collected will be handles following the most strict Good Clinical Practice (GCPs) and privacy norms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer who underwent radical prostatectomy;
* Adult patients > 18 years
* Ability to read and sign the informed consent

Exclusion Criteria:

* Patients < 18 years
* mental or physical disability that may prevent the patient from satisfying the requirements of the protocol
* Inability to read and sign the informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of prostate cancer who need to undergo radical prostatectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 1784 (Actual)
Dates: Start 2004-04-08 (Actual); Primary Completion 2025-02-13 (Estimated); Study Completion 2025-02-13 (Estimated)

PRIMARY OUTCOMES:
Early Urinary continence recovery | 6 months after the intervention/procedure/surgery
  Continence recovery evaluated with the International Consultation on Incontinence questionnaire - short form (ICIQ-SF), International Prostatic Symptoms Score (IPSS) questionnaires
Early Erectile function recovery | 6 months after the intervention/procedure/surgery
  Erectile function recovery evaluated with the International Index of Erectile Function (IIEF) questionnaire
Prostate-specific antigen (PSA) persistence or biochemical recurrence | 6 months and every year after the intervention/procedure/surgery up to 10 years
  Serum PSA levels, conventional imaging

SECONDARY OUTCOMES:
Urinary continence recovery | every year after the intervention/procedure/surgery up to 10 years
  Continence recovery evaluated with the International Consultation on Incontinence
Erectile function recovery | every year after the intervention/procedure/surgery up to 10 years
  Erectile function recovery evaluated with the International Index of Erectile Function (IIEF)

CONTACTS AND LOCATIONS:
Locations (1):
- Francesco Montorsi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No